CLINICAL TRIAL: NCT03651544
Title: An Open Study of the Safety, Reactogenicity and Immunogenicity of the GamFluVac Vector Vaccine Against Influenza A in Healthy Volunteers in 3 Groups With a Dose Escalation
Brief Title: The Study of the Safety, Reactogenicity and Immunogenicity of the GamFluVac
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 03-GamFluVac-2018
Record Dates: First submitted 2018-08-24; First posted 2018-08-29 (Actual); Last update posted 2019-03-15 (Actual); Status verified 2018-07

CONDITIONS: Influenza A Virus Infection; Influenza A; Influenza Epidemic; Influenza H5N1
Keywords: influenza; vaccine; vector vaccine
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Intervention Model Description: Taking into account the fact that the drug is being studied for the first time with the participation of people, initially 5 volunteers will be hospitalized, who will receive the study drug at a dose of 1. If the safety of the drug is confirmed by the results of observation on the 7th day of the study, the study will continue with the participation of 7 more volunteers in this dosing group.
  Further, according to a similar scheme (each time after an interim safety assessment on day 7), volunteers receiving the drug at a dose 2 and dose 3 will be included in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (GamFluVac dose1) (Experimental): The total number of recombinant pseudo-adenoviral particles (2.5 ± 1.25) x 1010 VP/dose.
  Interventions: Biological: GamFluVac
- Group 2 (GamFluVac dose2) (Experimental): Total amount of recombinant pseudo-adenoviral particles (1.0 ± 0.5) x 1011 VP/dose
  Interventions: Biological: GamFluVac
- Group 3 (GamFluVac dose3) (Experimental): The total number of recombinant pseudo-adenoviral particles (2.5 ± 1.25) × 1011 VP/dose
  Interventions: Biological: GamFluVac

INTERVENTIONS:
Biological: GamFluVac — 1 dose (0,5 ml)

SUMMARY:
The present clinical phase I study designed to examine the safety, reactogenicity and immunogenicity of the medicinal product - Vaccine vector against influenza A - in healthy volunteers after a single dose in the three groups with dose escalation.

DETAILED DESCRIPTION:
According to the results of the screening of volunteers who signed the informed consent Form, a sequential set of three groups of volunteers with different doses of the drug, the total number of volunteers who received the drug will be at least 36 people.

Given the fact that the drug is investigated for the first time with the participation of the people, will initially be admitted to hospital on 5 volunteers who will receive the investigational drug in the 1 dose The total number of recombinant pseudo-adenoviral particles (2.5 ± 1.25) x 10*10 VP/dose). If the safety of the drug is confirmed by the results of observation on the 7th day of the study, the study will continue with the participation of 7 more volunteers in this dosing group.

Further, according to a similar scheme (each time after an interim safety assessment on day 7), the study will include volunteers receiving the drug at a dose of 0.5 ml (Total amount of recombinant pseudo-adenoviral particles (1.0 ± 0.5) x 1011 VP/dose), particles/dose and 0.5 ml, -The total number of recombinant pseudo-adenoviral particles (2.5 ± 1.25) × 1011 VP/dose .

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged 18 to 55 years old.
* Written informed consent.
* consent to the use of effective contraceptive methods throughout the study period *

  * using one of the following methods: abstinence, condoms (male or female with or without spermicide), diaphragm or cervical cap with spermicide, intrauterine device
* body mass index (BMI) from 18.5 to 30.
* absence of acute infectious diseases or exacerbation of chronic infections at the time of vaccination and 7 days before vaccination;
* absence of allergic diseases of a serious degree (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum sickness)
* absence of strong post-vaccination reactions or post-vaccination complications for previous use of immunobiological drugs;
* absence of pathology from the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system, musculoskeletal system, genitourinary and endocrine systems, which may influence the evaluation of the results of the study, in the anamnesis and also according to the screening examination data;
* negative pregnancy test (for fertile women);
* negative tests for HIV, hepatitis B and C, syphilis;
* negative urine test for traces of drugs;
* negative test for alcohol content in the exhaled air;
* absence of malignant blood diseases;
* absence of malignant neoplasms;
* indicators of the total blood test at the screening not higher/lower than 1.1 x LLN/ULN (upper/lower limit of the normal reference range) *;

  * normal reference values of the laboratory performing the studies must be provided before the volunteer screening begins
* according to the biochemical blood test at the screening: the level of urea, creatinine, alanine aminotransferase, aspartate aminotransferase, glucose, creatine phosphokinase, total protein, bilirubin, glucose, LDH, alkaline phosphatase, LDL / HDL / VLDL - no higher/lower 1.1 X LLN/ULN (upper/lower limit of the normal reference range), total cholesterol level from 3,6 mmol/l to 7,8 mmol/l;
* no changes in myocardium of inflammatory or dystrophic nature according to ECG results at screening;
* lack of vaccination against influenza within 6 months before the start of the study (including during participation in other clinical trials).

Exclusion criteria

* participation of a volunteer in any other study in the last 90 days;
* any vaccination in the last 30 days;
* vaccination against influenza within 6 months before the start of the study (including during participation in other clinical trials).
* symptoms of respiratory illness in the last 3 days;
* recent frequent nasal bleeding (> 5 last year);
* chronic rhinitis, the presence of defects of the nasal septum, polyps of the nose or other significant anomalies;
* surgical operations or a history of nasal trauma for 6 months.
* treatment with steroids in the last 10 days;
* administration of immunoglobulins or other blood products for the last 3 months;
* taking immunosuppressive drugs and / or immunomodulators within 6 months before the start of the study;
* regular past or current use of narcotic drugs;
* pregnancy or breastfeeding;
* systolic blood pressure less than 100 mmHg or higher than 139 mmHg; diastolic blood pressure less than 60 mmHg. or above 90 mmHg; the heart rate is less than 60 beats per minute or more than 90 beats per minute;
* exacerbation of allergic diseases, the presence of anaphylactic reactions or angioedema in medical history;
* hypersensitivity or allergic reactions to the administration of any vaccine in medical history;
* allergic reactions to vaccine components;
* diabetes mellitus or other forms of impaired glucose tolerance;
* the presence of a concomitant disease that may influence the evaluation of the results of the study: active forms of tuberculosis, chronic liver and kidney diseases, severe thyroid dysfunction and other endocrine system diseases (diabetes mellitus), severe diseases of hematopoietic system, epilepsy and other CNS diseases, myocardial infarction, myocarditis, endocarditis, pericarditis, coronary heart disease, autoimmune pathology, serious chronic diseases requiring a hospitalisation;
* donor blood donation (450 ml and more blood or plasma) less than 2 months before the start of the study;
* taking a history of more than 5 units of alcohol (equal 0.25 liters of ethanol) per week;
* smoking: more than 10 cigarettes a day;
* planned hospitalization and / or surgical intervention during the study period, and 4 weeks before the expected date of vaccination.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-10-15 (Actual); Primary Completion 2018-12-24 (Actual); Study Completion 2019-03-14 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | Through the whole study, an average of 28 days
  Determination of Number of Participants With Adverse Events

SECONDARY OUTCOMES:
Assessment of antigen-specific cell-mediated immune response | at days 0 and 7
  determination of specific T-cell- mediated response vs. baseline values
Antibody levels a measured by an enzyme-linked immunosorbent assay (ELISA) | at days 0 and 28
  Determination of antibody levels measured by an ELISA vs. baseline values

CONTACTS AND LOCATIONS:
Overall Officials: Irina Gagarina, MD, PhD, Principal Investigator — Federal state budgetary institution " Main military clinical hospital named after academician N. N. Burdenko " of the Ministry of Defence of the Russian Federation
Locations (1):
- Federal state budgetary institution " Main military clinical hospital named after academician N. N. Burdenko " of the Ministry of Defence of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: Undecided